CLINICAL TRIAL: NCT03131973
Title: Effects of Concomitant Administration of BMS-986195 on the Single-dose Pharmacokinetics of Methotrexate and Probe Substrates for Cytochrome P450 1A2, 2C8, 2C9, 2C19, 3A4, Organic Anion Transporter Polypeptide 1B1 and P-glycoprotein in Healthy Participants
Brief Title: Effects of Concomitant Administration of BMS-986195 on Methotrexate, Caffeine, Montelukast, Flurbiprofen, Omeprazole, Midazolam, Digoxin, and Pravastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IM014-013
Record Dates: First submitted 2017-04-25; First posted 2017-04-27 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — branebrutinib; Methotrexate; Leucovorin; Caffeine; montelukast; Flurbiprofen; Omeprazole; Midazolam; Digoxin; Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Methotrexate (Experimental): Methotrexate single oral dose followed by leucovorin single oral dose on specified days followed by BMS-986195 coadministered with methotrexate single oral dose followed by leucovorin single oral dose on specified days
  Interventions: Drug: BMS-986195; Drug: Methotrexate; Drug: Leucovorin
- Cytochrome P450 and Transporter Substrates (Experimental): Caffeine, montelukast, flurbiprofen, omeprazole, midazolam, digoxin, and pravastatin single oral dose on specified days, BMS-986195 multiple oral dose administration on specified days, and BMS-986195 coadministered with caffeine, montelukast, flurbiprofen, omeprazole, midazolam, digoxin, and pravastatin single oral dose on specified days.
  Interventions: Drug: BMS-986195; Drug: Caffeine; Drug: Montelukast; Drug: Flurbiprofen; Drug: Omeprazole; Drug: Midazolam; Drug: Digoxin; Drug: Pravastatin

INTERVENTIONS:
Drug: BMS-986195 — Specified dose on specified days
Drug: Methotrexate — Specified dose on specified days
  Arms: Methotrexate
Drug: Leucovorin — Specified dose on specified days
  Arms: Methotrexate
Drug: Caffeine — Specified dose on specified days
  Arms: Cytochrome P450 and Transporter Substrates
Drug: Montelukast — Specified dose on specified days
  Arms: Cytochrome P450 and Transporter Substrates
Drug: Flurbiprofen — Specified dose on specified days
  Arms: Cytochrome P450 and Transporter Substrates
Drug: Omeprazole — Specified dose on specified days
  Arms: Cytochrome P450 and Transporter Substrates
Drug: Midazolam — Specified dose on specified days
  Arms: Cytochrome P450 and Transporter Substrates
Drug: Digoxin — Specified dose on specified days
  Arms: Cytochrome P450 and Transporter Substrates
Drug: Pravastatin — Specified dose on specified days
  Arms: Cytochrome P450 and Transporter Substrates

SUMMARY:
Drug-drug interaction study in healthy men and women not of childbearing potential. Assess the effect of BMS-986195 on the pharmacokinetics of methotrexate, caffeine, montelukast, flurbiprofen, omeprazole, midazolam, digoxin, and pravastatin. Collect data on safety of BMS-986195 and methotrexate, caffeine, montelukast, flurbiprofen, omeprazole, midazolam, digoxin, and pravastatin. Collect data on multiple-dose pharmacodynamics of BMS-986195.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female (not of childbearing potential) participants as determined by medical and surgical history and assessments
* Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive
* Normal kidney function at screening

Exclusion Criteria:

* History of chronic headaches (eg, migraines, cluster headaches), defined as occurring 15 days or more a month, over the previous 3 months
* History of headaches related to caffeine withdrawal, including energy drinks
* History of syncope, orthostatic instability, or recurrent dizziness

Other protocol defined inclusion and exclusion criteria could apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-05-13 (Actual); Primary Completion 2017-11-05 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 26 days
  Measured by plasma concentrations
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) | Up to 26 days
  Measured by plasma concentrations
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Up to 26 days
  Measured by plasma concentrations

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 28 days
  Measured by investigator assessment
Number of participants with serious adverse events | Up to 45 days
  Measured by investigator assessment
Number of participants with adverse events leading to discontinuation | Up to 28 days
  Measured by investigator assessment
Number of participants with clinical laboratory test abnormalities | Up to 28 days
Number of participants with vital sign measurement abnormalities | Up to 28 days
Number of participants with electrocardiogram abnormalities | Up to 28 days
Number of participants with physical examination abnormalities | Up to 28 days
Number of participants with marked abnormalities in clinical laboratory test results | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Development, LP, Austin, Texas, United States

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/